CLINICAL TRIAL: NCT04777851
Title: A Phase III, Multicenter, Randomized, Open-label Trial to Evaluate the Safety and Efficacy of Systemic Therapy With Regorafenib and Pembrolizumab Versus Locoregional Therapy With Transarterial Chemoembolization or Transarterial Radioembolization, for the First-line Treatment of Intermediate-stage Hepatocellular Carcinoma With Beyond Up-to-7 Criteria
Brief Title: Regorafenib-pembrolizumab vs. TACE/TARE in Intermediate Stage HCC Beyond Up-to-7
Acronym: REPLACE
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Translational Research in Oncology (Other)
Collaborators: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TRIO041; EU CT # 2022-501969-42-00 (Other: European Medicines Agency (EMA))
Record Dates: First submitted 2021-02-25; First posted 2021-03-02 (Actual); Last update posted 2025-05-15 (Actual); Status verified 2025-05

CONDITIONS: Carcinoma, Hepatocellular
Keywords: Hepatocellular Carcinoma; Hepatoma; Liver Cancer, Adult; Liver Cell Carcinoma; Liver Cell Carcinoma, Adult
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — regorafenib; pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Regorafenib + Pembrolizumab (Experimental): Investigational arm: regorafenib at a dose of 90 mg orally once per day (on days 1 to 21 of a 28-day cycle), in combination with pembrolizumab 400 mg using a 30-minute intravenous infusion, on day 1 of a 6-week cycle.
  Interventions: Drug: Regorafenib in combination with pembrolizumab
- Loco-regional therapy (Active Comparator): Control arm: Patients will be treated with TACE or TARE "on-demand" according to site's standard of practice.
  Interventions: Procedure: Loco-regional therapy

INTERVENTIONS:
Drug: Regorafenib in combination with pembrolizumab — Randomized patients will receive regorafenib at a dose of 90 mg per day by mouth on days 1 to 21 of a 28-day cycle, in combination with pembrolizumab 400 mg using a 30-minute intravenous infusion, on day 1 (D1) of a 6-week cycle.
  Other Names: Stivarga® (regorafenib); Keytruda® (pembrolizumab)
  Arms: Regorafenib + Pembrolizumab
Procedure: Loco-regional therapy — Patients will be treated with TACE or TARE "on-demand" according to site's standard of practice.
  Other Names: Convention transarterial chemoembolization (cTACE); Drug-eluting bead transarterial chemoembolization (DEB-TACE); Transarterial Chemoembolization (TACE); Transarterial radioembolization (TARE)
  Arms: Loco-regional therapy

SUMMARY:
REPLACE is a phase III, multicenter, randomized, open-label trial to evaluate the efficacy and safety of regorafenib and pembrolizumab (Rego-Pembro) versus transarterial chemoembolization (TACE) or transarterial radioembolization (TARE) for the first-line treatment of hepatocellular carcinoma (HCC or liver cancer). Approximately 496 patients in around 80 clinical sites worldwide will be randomized to receive either:

* Investigational arm: Regorafenib in combination with pembrolizumab
* Control arm: Transarterial chemoembolization (TACE) or transarterial radioembolization (TARE)

In both arms, patients will receive trial treatment until progressive disease, unacceptable toxicity, deterioration of patient's condition that warrants permanent trial treatment discontinuation or other treatment discontinuation criteria is met. After trial treatment discontinuation, subsequent treatment will be administered according to the Investigator's clinical judgment.

DETAILED DESCRIPTION:
REPLACE is a phase III, multicenter, randomized, open-label trial to evaluate the efficacy and safety of systemic therapy with Rego-Pembro versus loco-regional therapy with TACE or TARE, for the first-line treatment of intermediate-stage HCC with beyond up-to-7 criteria. Approximately 496 patients (~248 in each arm) from approximately 80 sites will be randomized in order to power the trial efficiently to measure a clinically meaningful improvement for the primary endpoint, PFS according to mRECIST based on the Investigator´s assessment.

The trial will include patients who have been diagnosed with intermediate-stage HCC by biopsy, cytology or diagnostic imaging, such as dynamic computed tomography (CT) or magnetic resonance imaging (MRI), according to the criteria of the American Association for the Study of Liver Diseases (AASLD). Patients should have at least one measurable lesion per RECIST 1.1, disease not amenable to curative treatment but amenable to loco-regional therapy with TACE (cTACE or DEB-TACE) or TARE, ECOG PS 0-1, Child-Pugh class A, and beyond up-to-7 criteria.

The trial will include the following phases:

* Screening
* Treatment
* Follow-up

Randomized patients will receive either:

Investigational arm (Arm A):

-Regorafenib at a dose of 90 mg orally q.d. on days 1 to 21 of a 4-week cycle.

In combination with:

-Pembrolizumab 400 mg using a 30-minutes i.v. infusion, on day 1 (D1) of a 6-week cycle.

Control arm (Arm B):

-Patients will be treated with TACE or TARE "on-demand" according to site's standard, with the goal of controlling all known liver lesions.

In both arms, patients will receive trial treatment (Rego-Pembro or TACE/TARE) until PD per mRECIST, unacceptable toxicity, deterioration of patient's condition that warrants permanent trial treatment discontinuation or other treatment discontinuation criteria are met.

ELIGIBILITY:
Inclusion Criteria:

* Signed and dated Patient Informed Consent Form (PICF)
* ≥ 18 years-old at the time of PICF signature
* Confirmed diagnosis of HCC
* Intermediate-stage HCC, defined as follows:

  * Multinodular HCC localized to the liver
  * No evidence of MVI or EHS
  * Not amenable to curative treatment
  * Child-Pugh Class A
  * ECOG PS 0 or 1
  * ALBI grade 1 or 2
* Beyond up-to-seven criteria
* Disease amenable to TACE or TARE and no contradiction to intra-arterial treatment
* Measurable disease by CT or MRI as per RECIST 1.1
* No prior systemic therapy or loco-regional therapy for HCC
* Adequate hematologic and organ function
* Willing and able to comply with scheduled visits, treatment plans, laboratory tests and other trial procedures
* Women of childbearing potential (CBP) must have confirmed negative serum pregnancy test
* Use of highly-effective contraceptive methods in women of CBP and men
* Patients with hepatitis C virus (HCV) or hepatitis B virus (HBV) infection are eligible if they meet criteria as defined within the protocol

Exclusion Criteria:

* No measurable tumor of a diffuse infiltrative HCC type.
* Fibrolamellar HCC, sarcomatoid HCC or mixed hepatocellular/ cholangiocarcinoma subtypes.
* Clinically meaningful ascites.
* Prior treatment with regorafenib, a PD-1, PD-L1/PD-L2, or cytotoxic T lymphocyte associated protein 4 (CTLA-4) inhibitors, or any other antibody or drug specifically targeting T-cell co-stimulation or checkpoint pathways.
* Major surgical procedure, open biopsy, or significant traumatic injury ≤28 days prior to randomization.
* Active autoimmune disease or history of autoimmune disease that might recur, which may affect vital organ function or require immune suppressive treatment including systemic corticosteroids.
* Requirement of systemic treatment with either corticosteroids or other immunosuppressive medications ≤ 14 days prior to randomization.
* Interstitial lung disease, non-infectious pneumonitis or uncontrolled lung diseases including pulmonary fibrosis, or clinically significant acute lung diseases.
* Cardiovascular conditions as defined within the protocol.
* Patient has a concurrent invasive malignancy or a prior invasive malignancy whose treatment was completed ≤ 2 years before randomization.
* Persistent proteinuria of NCI-CTCAE v5.0 Grade 3.
* Pregnant or breast-feeding (lactating) women or women who plan to become pregnant or breast-feed during the trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 496 (Estimated)
Dates: Start 2023-10-11 (Actual); Primary Completion 2026-02-28 (Estimated); Study Completion 2026-02-28 (Estimated)

PRIMARY OUTCOMES:
Progression-free Survival (PFS) Assessed by the Investigator as per Modified Response Evaluation Criteria in Solid Tumors (mRECIST) for HCC | up to 3.5 years
  PFS, defined as the time (in months) from the date of randomization until the date of progressive disease (PD) or death due to any cause, whichever occurs first. PD will be assessed locally by the Investigator using mRECIST.

SECONDARY OUTCOMES:
Progression-free Survival (PFS) Assessed by the Investigator as per Response Evaluation Criteria in Solid Tumors (RECIST) Version 1.1 | up to 3.5 years
  PFS, defined as the time (in months) from the date of randomization until the date of progressive disease (PD) or death due to any cause, whichever occurs first. PD will be assessed locally by the Investigator using RECIST 1.1.
Progression-free Survival (PFS) Assessed by Blinded Independent Central Review (BICR) as per Modified Response Evaluation Criteria in Solid Tumors (mRECIST) and RECIST Version 1.1 | up to 3.5 years
  PFS, defined as the time (in months) from the date of randomization until the date of PD or death due to any cause, whichever occurs first. PD will be assessed by BICR using, independently, mRECIST and RECIST 1.1.
Overall Survival (OS) of Intermediate-Stage HCC (Rego-Pembro versus Loco-regional Therapy) | up to 3.5 years
  OS, defined as the time (in months) from the date of randomization until the date of death due to any cause.
Overall Response Rate (ORR) Assessed by Investigator and Blinded Independent Central Review (BICR) as per Modified Response Evaluation Criteria in Solid Tumors (mRECIST) and RECIST Version 1.1 | up to 3.5 years
  ORR, defined as the proportion of patients who have a complete response (CR) or partial response (PR) according to RECIST v.1.1 and mRECIST, based on the Investigator's and BICR assessment.
Time to unTACEable Progression (TTUP) | up to 3.5 years
  To evaluate the two treatment arms (rego-pembro versus loco-regional therapy) with respect to TTUP. TTUP, defined as the time (in months) from the date of randomization until any of the following criteria are met:
  * Factors related to liver function:
    * Decompensated cirrhosis (Child-Pugh class B score > 8), including jaundice, clinical hepatic encephalopathy, and refractory ascites and/or hepatorenal syndrome
    * Impaired portal-vein blood flow (portal-vein thrombus, hepatofugal blood flow)
    * ECOG PS ≥ 2 Note: transient post-TACE/TARE impairment of liver function of Child-Pugh class B score > 8, that return to pre-TACE/TARE values within 4 weeks of the TACE/TARE session will not qualify as TTUP.
  * Factors related to HCC:
    * Failure of the treated nodule to achieve Stable Disease (SD), PR or CR by mRECIST
    * Malignant portal vein thrombosis
    * Marcovascular invasion (MVI) or Extra-hepatic Spread (EHS)
Duration of Response (DOR) of Rego-Pembro Versus Loco-regional Therapy | up to 3.5 years
  To evaluate the two treatment arms with respect to DOR. DOR, defined as the time (in months) from first documentation of response (PR or CR) to PD or death, based on Investigator's assessment or death from any cause, in patients who had a best overall response of CR or PR.
Number of Patients with Adverse Events as Assessed by the National Cancer Institute Common Terminology Criteria of Adverse Events (NCI-CTCAE) Version 5 | up to 3.5 years
  The NCI-CTCAE is a descriptive terminology which can be utilized for Adverse Event (AE) reporting. A grading scale is provided for each AE term with unique clinical descriptions of severity based on this general guideline: Grade 1 (mild) to 5 (death). AEs will be tabulated by treatment arm, system organ class, preferred term, severity, and relationship to treatment.
Change from Baseline in the Physical Functioning Sub-scale Score and Global Health Status/Quality of Life Scale Score as assessed by European Organization for Research and Treatment of Cancer's Core Quality of Life Questionnaire (EORTC QLQ-C30) | up to 3.5 years
  To evaluate the patient reported outcomes in the two treatment arms (rego-pembro versus loco-regional therapy) as assessed by EORTC QLQ C30. EORTC QLQ C30 is a quality-of-life questionnaire to assess patients' physical, psychological and social functions. The questionnaire is composed of functional scales (physical, role, cognitive, emotional, social), symptom scales (fatigue, pain, and nausea and vomiting), global health status and quality of life scale, also several single-item symptom measures (scaling of items: 1 = Not at all to 4 = Very much; 1 = Very poor to 7 = Excellent). Scores range from 0 to 100, with a high score representing a better health-related quality of life.
Change from Baseline in Health-related Quality of Life in Hepatocellular Carcinoma as Assessed by European Organization for Research and Treatment of Cancer's Quality of Life Questionnaire for HCC (EORTC QLQ-HCC18) | up to 3.5 years
  To evaluate patient reported outcomes in the two treatment arms (rego-pembro versus loco-regional therapy) as assessed by EORTC QLQ-HCC18. EORTC QLQ-HCC18 is an 18-question module specifically to assess symptom burden and impact on health-related quality of life measuring HCC-specific symptoms. The instrument is an 18-item scale, and scores are based on a 4-point Likert scale (with 1 = 'not at all' to 4 = 'very much'); scaled scores range from 0-100 with a higher score indicating worse symptoms.
Change from Baseline in Health-Related Quality of Life as Assessed by the EuroQol's 5-level EQ-5D Health Questionnaire (EQ-5D-5L) | up to 3.5 years
  To evaluate patient reported outcomes for health-related quality of life in the two treatment arms (rego-pembro versus loco-regional therapy) as assessed by health questionnaire EQ-5D-5L. Each dimension (Mobility, Self-care, Usual activities, Pain & discomfort, Anxiety & depression) in the EQ-5D-5L has five response levels: no problems (Level 1); slight; moderate; severe; and extreme problems (Level 5). There are 3,125 possible health states defined by combining one level from each dimension, ranging from 11111 (full health) to 55555 (worst health).

CONTACTS AND LOCATIONS:
Overall Officials: Peter R Galle, MD, Study Chair — University Medical Center, Mainz, Germany; Richard S Finn, MD, Study Chair — UCLA Department of Medicine, Division of Hematology-Oncology
Locations (26):
- UCLA Santa Monica Hematology Oncology, Santa Monica, California, United States
- Belgium (2):
  - UCL SAINT LUC - UC Louvain, Brussels
  - Antwerp University Hospital, Edegem
- France (3):
  - CHU Amiens-Picardie, Amiens
  - Hôpital Beaujon - APHP, Clichy
  - Hôpital Henri Mondor, Créteil
- Georgia (2):
  - JSC VIANI Batumi Referral Hospital, Batumi
  - Israel-Georgian Medical Research Clinic Healthycore, Tbilisi
- Universitätsmedizin: Medizinische Klinik und Poliklinik I, Mainz, Germany
- Humanity and Health Clinical Trial Center, Hong Kong, Hong Kong
- Ospedale Garibaldi Nesima, Catania, Italy
- Romania (3):
  - Institutul Clinic Fundeni, Bucharest
  - Regional Institute of Gastroenterology and Hepatology "Dr Octavian Fodor", Cluj-Napoca
  - Center of Oncology Euroclinic Victoria Hospital, Iași
- Serbia (2):
  - Clinic for Digestive Surgery, University Clinical Center of Serbia, Belgrade
  - Institue of Oncology Vojvodine Sremska Kamenica (Oncology Institute of Volvodina), Kamenitz
- South Korea (3):
  - Inje University Haeundae Paik Hospital, Busan
  - Cha Bundang Medical Center, Seongnam-si
  - Severance Hospital, Yonsei University Health System, Seoul
- Spain (2):
  - Hospital Universitario La Paz, Madrid
  - Hospital Universitario Miguel Servet, Zaragoza
- Taiwan (2):
  - National Taiwan University Hospital, Taipei
  - Chang Gung Memorial Hospital - Linkou, Taoyuan District
- Turkey (Türkiye) (3):
  - Gülhane Eğitim ve Araştırma Hastanesi, Ankara
  - Gazi University MF, Ankara
  - Koc University Hospital, Istanbul